CLINICAL TRIAL: NCT00286156
Title: Pilot Study of Rapamycin as Treatment for Autosomal Dominant Polycystic Kidney Disease
Brief Title: Pilot Study of Rapamycin as Treatment for Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 7736
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2014-03

CONDITIONS: Polycystic Kidney Diseases
Keywords: ADPKD
MeSH Terms: conditions — Polycystic Kidney Diseases; Polycystic Kidney, Autosomal Dominant | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Arm 1 Rapamune dose 2-6mg aimed at maintaining trough levels 5-8 ng/ml
  Interventions: Drug: Rapamune
- 2 (Experimental): Arm 2 Rapamune dose 2-6 mg aimed at maintaining trough levels of 2-5ng/ml
  Interventions: Drug: Rapamune
- 3 (No Intervention): Standard Care

INTERVENTIONS:
Drug: Rapamune — Group 1- doses of Rapamune aimed at maintaining trough levels 5-8ng/ml Group 2 - doses of Rapamune aimed at maintaining trough levels 2-5ng/ml Group 3- Standard Care
  Other Names: Rapamycin
  Arms: 1; 2

SUMMARY:
This study is a prospective, randomized, open-label, pilot clinical trial designed to compare the effects of an agent that has antiproliferative (1,2), antiangiogenesis (3),and tumor-progression blocking capabilities (4), namely, rapamycin (Rapamune®), in the treatment of autosomal-dominant polycystic kidney disease (ADPKD).

Up to this time, only generic renal disease treatments for ADPKD have been in use, such as the treatment of hypertension, urinary tract infections, renal stones, renal call carcinomas, and replacement therapy with dialysis and/or renal transplantation. The fundamental aberrations in ADPKD are proliferation of cyst-forming tubuloepithelial cells, secretion of cytokine-rich fluid into those cysts, and progressive cyst expansion and release of inflammatory mediators that injure surrounding normal renal tissue. Consequently, therapy directed specifically at blocking the proliferation of tubuloepithelial cells and their tendency to malignant transformation, as well as impeding their blood supply, should have obvious merit.

General Procedures:

In Group I participants will have an iothalamate glomerular filtration rate (GFR) equal to or greater than 60 ml/min/1.73 m2, and in Group II participants will have a GFR less than 25-59 ml/min/1.73 m2. Both males and females with ADPKD who volunteer and qualify, will be randomly and prospectively assigned to treatment with rapamycin at either a high or low trough blood level or to standard care (each 1/3 of enrolled patients) for one year. The two treatment groups will receive rapamycin doses aimed at maintaining the 20- to 24-hour trough blood levels at either 2 to 5 ng/mL (low-dose), or greater than 5 to 8 ng/mL (high-dose). These trough levels are in the lower range of levels used when treating renal transplant recipients in whom trough levels are typically maintained between 5 and 15 ng/mL.

DETAILED DESCRIPTION:
This study is a prospective, randomized,open label, pilot clinical trial designed to compare the effects of an agent that has antiproliferative (1,2), antiangiogenesis (3),and tumor-progression blocking capabilities (4), namely, rapamycin (Rapamune®), in the treatment of autosomal-dominant polycystic kidney disease (ADPKD).

Up to this time, only generic renal disease treatments for ADPKD have been in use, such as the treatment of hypertension, urinary tract infections, renal stones, renal call carcinomas, and replacement therapy with dialysis and/or renal transplantation. The fundamental aberrations in ADPKD are proliferation of cyst-forming tubuloepithelial cells, secretion of cytokine-rich fluid into those cysts, and progressive cyst expansion and release of inflammatory mediators that injure surrounding normal renal tissue. Consequently, therapy directed specifically at blocking the proliferation of tubuloepithelial cells and their tendency to malignant transformation, as well as impeding their blood supply, should have obvious merit.

General Procedures:

In Group I participants will have an iothalamate glomerular filtration rate (GFR) equal to or greater than 60 ml/min/1.73 m2, and in Group II participants will have a GFR less than 25-59 ml/min/1.73 m2. Both males and females with ADPKD who volunteer and qualify, will be randomly and prospectively assigned to treatment with rapamycin at either a high or low trough blood level or to standard care (each 1/3 of enrolled patients) for one year. The two treatment groups will receive rapamycin doses aimed at maintaining the 20- to 24-hour trough blood levels at either 2 to 5 ng/mL (low-dose), or greater than 5 to 8 ng/mL (high-dose). These trough levels are in the lower range of levels used when treating renal transplant recipients in whom trough levels are typically maintained between 5 and 15 ng/mL.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD
* > 18 y.o. GFR greater than or equal to 25. Willingness to be randomized to any treatment group Willingness to follow protocol requirements-frequent testing and follow-up required at Cleveland Clinic(Cleveland, OH) signed informed consent Willingness to use birth control(male and female)

Exclusion Criteria:

* Pregnancy
* post partum
* lactating
* system illness with renal involvement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2012-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E. Braun, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic- main campus, Cleveland, Ohio, United States

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Rapamycin Dose (STD): Arm 1 Rapamune dose 2-6mg aimed at maintaining trough levels 5-8 ng/ml
  Rapamycin: Group 1- doses of Rapamune aimed at maintaining trough levels 5-8ng/ml
- Low Dose Rapamycin (LD): Arm 2 Rapamune dose 2-6 mg aimed at maintaining trough levels of 2-5ng/ml
  Rapamycin: Group 2 - doses of Rapamune aimed at maintaining trough levels 2-5ng/ml
- Standard Care: Standard Care: fluid intake primarily water of 2500-3000ml/24hrs, low sodium diet of 2300mg/24 hrs, caffeine avoidance, control of hypertension
Period: Overall Study
Arm/Group | Standard Rapamycin Dose (STD) | Low Dose Rapamycin (LD) | Standard Care
Started | 10 | 10 | 10
Completed | 8 | 9 | 9
Not Completed | 2 | 1 | 1
Not completed — Missed 12 month visit | 0 | 0 | 1
Not completed — AE: pulmonary embolus | 0 | 1 | 0
Not completed — AE: nephrotic-range proteinuruia | 1 | 0 | 0
Not completed — AE: pneumonia | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Rapamycin Dose (STD) | Low Dose Rapamycin (LD) | Standard Care | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (15.0) | 44.9 (8.6) | 49.4 (11.0) | 49.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 13
  Male | 5 | 5 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 10 | 9 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Baseline characteristics and risk factors [Number; unit: participants] — ADPKD, autosomal dominant polycystic kidney disease; iGFR, 125I-iothalamate GFR; TKV, total kidney volume; Hypertension is a BP >= 140/90 mmHg before 35 years old; family history of ESRD occurs from ADPKD before 56 years old
  participants
    Hypertension | 3 | 3 | 5 | 11
    Family history of ESRD | 4 | 8 | 7 | 19
    Initial iGFR 25-59 ml/min per 1.73 m^2 | 3 | 4 | 2 | 9
    Initial TKV>1500ml | 6 | 7 | 6 | 19
    Initial height-adjusted TKV>=600ml/m | 6 | 8 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in GFR From Baseline to 12 Months
Description: GFR (glomerular filtration rate) was measured by iothalamate. GFR is a key indicator of renal function.
Time Frame: From baseline to 12 months
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Standard Rapamycin Dose (STD) | Low Dose Rapamycin (LD) | Standard Care
Number analyzed (Participants) | 8 | 9 | 9
ml/min/1.73m^2
  Baseline iGFR | 72.8 (25.7) | 70.3 (27.0) | 73.1 (20.3)
  12 month iGFR | 74.4 (34.4) | 78.0 (35.0) | 61.9 (15.6)
  Change in iGFR | 1.6 (12.1) | 7.7 (12.5) | -11.2 (9.1)
Statistical Analysis 1: Comparison: Standard Rapamycin Dose (STD) vs Low Dose Rapamycin (LD) vs Standard Care; Null hypothesis: no difference between groups in iGFR; Test type: Superiority or Other; p < 0.01, ANOVA — Pairwise comparisons adjusted for multiple testing (Tukey)

2. Secondary Outcome: Change in Total Kidney Volume as Measured by 3D-CT From Baseline to 12 Months
Description: Total kidney volume measured by CT from baseline to 12 months
Time Frame: From baseline to 12 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Standard Rapamycin Dose (STD) | Low Dose Rapamycin (LD) | Standard Care
Number analyzed (Participants) | 8 | 9 | 9
ml
  Baseline TKV | 1454.1 (801.5) | 1919.1 (903.6) | 1907.1 (1126.8)
  12 month TKV | 1537 (864.3) | 2115.8 (1035.0) | 2059.8 (1236.0)
  Change in TKV | 82.9 (111.3) | 197.7 (201.2) | 152.7 (129.4)

ADVERSE EVENTS:
Arm/Group | Standard Rapamycin Dose (STD) | Low Dose Rapamycin (LD) | Standard Care
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 6/10 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Rapamycin Dose (STD) (N=10) | Low Dose Rapamycin (LD) (N=10) | Standard Care (N=10)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Patient had massive polycystic kidneys (about 7500ml) and there was compression of the right iliac vein/IVC with clot formation. This has been reported in the literature, so it is not necessarily related to drug.
nephrotic range proteinuria (Renal and urinary disorders) | 1 | 0 | 0 — Open renal biopsy showed FSGS. Primary glomerulopathies have been reported to be superimposed on underlying ADPKD.
Decrease visual acuity (Eye disorders) | 1 | 0 | 0 — Patient developed transient decrease in visual acuity. Neuro-ophthalmologist did not find any association with drug. Vision improved without specific treatment.
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 — Hypoglycemia associated with excessive beer consumption.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Rapamycin Dose (STD) (N=10) | Low Dose Rapamycin (LD) (N=10) | Standard Care (N=10)
Oral ulcerations (Immune system disorders) | 6 (6) | 2 (2) | 0 (0)
Nonserious infections (Infections and infestations) | 6 (6) | 2 (2) | 5 (5)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal symptoms (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Miscellaneous/other (General disorders) | 4 (7) | 2 (2) | 5 (7) — The problems in this group were minor, extremely varied and transient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes